CLINICAL TRIAL: NCT06057480
Title: A Prospective, Multicenter, Single-arm Study Examining the Assisted Programming Module (APM) in the Evoke Spinal Cord Stimulation (SCS) System to Program Patients With Chronic Pain of the Trunk and/or Limbs
Brief Title: APM in the Evoke SCS System to Program Patients With Chronic Pain of the Trunk and/or Limbs
Acronym: APM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D103684
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- APM (Experimental): Investigational programming software module, the Assisted Programming Module (APM)
  Interventions: Device: APM

INTERVENTIONS:
Device: APM — Investigational programming software module, the Assisted Programming Module (APM)

SUMMARY:
Study to evaluate the use of the Assisted Programming Module (APM) in the Evoke Spinal Cord Stimulation (SCS) System to program patients with chronic pain of the trunk and/or limbs.

ELIGIBILITY:
Inclusion Criteria:

* Subject has or is planning to undergo a temporary trial with Evoke System within the FDA approved indication.
* Subject is willing and capable of giving informed consent and able to comply with study-related requirements.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Evoked Compound Action Potentials (ECAPs) measured in µV by the Evoke SCS System | end of trial period; 1 month and 3 months post-implant
  Change in Evoked Compound Action Potentials (ECAPs) measured in µV by the Evoke SCS System
Change in programming parameters (e.g., stimulation frequency [Hz], pulse width [µs], amplitude [mA]) measured by the Evoke SCS System | end of trial period; 1 month and 3 months post-implant
  Change in programming parameters (e.g., stimulation frequency [Hz], pulse width [µs], amplitude [mA]) measured by the Evoke SCS System

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Pacific Research Institute, Santa Rosa, California
  - The Orthopaedic Institute, PA, Gainesville, Florida
  - Center for Clinical Research, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker DJ, Antony AB, Smith GL, Goree JH, Russo MA, Petersen EA, Vu CM, Verrills P, Gilmore C, Kapural L, Nanavati D, Karantonis DM, Pope JE. Next-Generation SCS Programming Platform: Enhancing ECAP Fidelity and Objectivity to Improve Patient Experience. Pain Ther. 2026 Jan 8. doi: 10.1007/s40122-025-00808-5. Online ahead of print. PMID 41505067